CLINICAL TRIAL: NCT06625632
Title: Effect of Kinesiotape on Emesis in Pregnant Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Soad Mansour Shawky El-Kholy, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005305
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Emesis Pregnancy
MeSH Terms: interventions — Antiemetics; Ondansetron; Vitamin B 6

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antiemetic drug + Vitamin B6 + Home care advice + Kinesiotaping (Experimental): It will be consisted of 25 pregnant women who will receive kinesiotaping (I band) for 5 days in addition to antiemetic drugs (ondansetron 4 mg, every 12 hours), vitamin B6 (50 mg, once daily), and home care advice.
  Interventions: Drug: Antiemetic Drug; Dietary Supplement: Vitamin B6; Other: Home care advice; Other: Kinesiotaping
- Antiemetic drug + Vitamin B6 + Home care advice (Active Comparator): It will be consisted of 25 pregnant women who will receive antiemetic drugs (ondansetron 4mg every 12 hours, vitamin B6 (50 mg, once daily), and home care advice only for 5 days.
  Interventions: Drug: Antiemetic Drug; Dietary Supplement: Vitamin B6; Other: Home care advice

INTERVENTIONS:
Drug: Antiemetic Drug — All participants in the two groups will receive antiemetic drugs (ondansetron 4 mg) every 12 hours, for 5 days.
  Other Names: Ondansetron 4 mg
Dietary Supplement: Vitamin B6 — All participants in the two groups will receive vitamin B6 (50 mg), once daily, for 5 days.
Other: Home care advice — All participants in both groups will be advised to eat small portions of food, drink plenty of liquids, and avoid fatty and fried foods. Additionally, they should steer clear of highly spiced foods, foods and beverages with strong odors, caffeine, and consume neither very hot nor very cold foods and liquids.
Other: Kinesiotaping — It will be applied for all participants in the experimental group only for 5 days. The participant will be asked to stand in erect position, her hands beside her body then applying the kinesiotape from origin (from top to bottom where the stomach is placed on the abdominal region) to insertion (alongside the gastric curvature) with tension 25% for 5 days.
  Arms: Antiemetic drug + Vitamin B6 + Home care advice + Kinesiotaping

SUMMARY:
This study will be conducted to investigate the effect of kinesiotaping on emesis in pregnant women.

DETAILED DESCRIPTION:
Emesis gravidarum (EG) is a common condition among pregnant women, with a prevalence of 12.5% worldwide. It has a significant impact on the body where the mother becomes very weak, the face is pale and the frequency of urination decreases drastically so, the body fluids are reduced, and blood becomes thick (hem concentration). This condition can slow down blood circulation so that oxygen and food supply to the tissues are also reduced which can cause tissue damage and endangers the health of the mother and her fetus. Also, EG known to reduce a woman's quality of life (QOL). It was reported that 80% of women with emesis have reduced QOL.

Women with EG fear from the use of the antiemetic drugs and the possible side effects such as drowsiness, sedation, arrhythmia, poor efficacy of pharmacological approach in the past leads to difficulty in the treatment of nausea and vomiting during pregnancy. Non- pharmacological option has been proposed to be effective in the treatment of EG and hyperemesis gravidarum. Such as hypnosis, acustimulation, tactile massage, psychotherapy, acupuncture and kinesiotape.

Kinesiotape is a drug-free and an elastic therapeutic tape used for treating various musculoskeletal problems such as injury, pain, and dysfunction and a variety of other disorders. The kinesiotaping was found to be effective in stimulation of large and small intestinal peristalsis.

Due to lack of previous studies that examined the effect of kinesiotape on EG. This raises the need of further studies in this issue which will give an insight about the efficacy of kinesiotape as a safe, non-invasive and inexpensive method used to alleviate nausea and vomiting during pregnancy. This will be of valuable benefits in medical service organization and increase body of knowledge of physical therapists in scientific field.

ELIGIBILITY:
Inclusion Criteria:

* Fifty pregnant women at 6th to 12th weeks of gestation diagnosed with mild to moderate nausea and vomiting.
* The diagnosis of EG is confirmed by Rhodes index.
* Their ages will be ranged from 20 to 35years old.
* Their body mass index will be less than 30 kg/m2.
* All of them are primigravida.

Exclusion Criteria:

* Digestive system diseases, inflammatory bowel disease, gastric ulcers and/or esophagitis.
* Twins or more.
* Obese women with BMI <30 kg/m2.
* Severe emesis or hyperemesis gravidarum.
* Risk of threatened or habitual abortion.
* Multi gravida.
* Thyroid or liver dysfunction.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2024-10-07 (Estimated); Primary Completion 2025-01-07 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | 24 hours
  It will be used for all participants in both groups pre and post-treatment to assess the severity of symptoms of emesis gravidarum. Patients will be asked on their first visit to grade the severity of their nausea over the past 24 hours (baseline scores) by marking an "X" corresponding to their perceived states on a 10-cm horizontal line, ranging from 0 no nausea to 10 nausea as bad as it could be. On the following 2 weeks of treatment, recordings of the severity of nausea will be made twice daily at noon and at bedtime.
Rhodes index | 24 hours
  It will be used for all participants in both groups pre and post-treatment to assess severity of nausea and vomiting for all participants in both groups before and after the study. Each woman will be asked to self-report questions such as length and episodes of nausea, number of vomits, number of retches, and volume of vomits on the 5-point scale with 1 indicating minimal or no symptom and 5 representing the worst symptom.
Pregnancy unique quantification of emesis (PUQE) | 24 hours
  It will be used for all participants in both groups pre and post-treatment to assess the symptoms of emesis gravidarum. This questionnaire contains three questions regarding the time-span of nausea, vomiting and retching respectively, as well as one question assessing the global psychological and physical quality of life (QOL). Each woman will be asked to choose the answer that suit the best of her situation for the last 24 hours. The PUQE score is calculated by adding the values from each category, and can range from a minimum of 1 to a maximum of 15, with higher scores indicating worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Azza Barmoud Nashed Kassab, PhD, Study Chair — Professor, Cairo university
Locations (1):
- Cairo University, Giza, Egypt